CLINICAL TRIAL: NCT03636568
Title: Early Fluid Restriction to Prevent Delayed Hyponatremia Following Pituitary Surgery
Brief Title: Hyponatremia Study (Delayed Hyponatremia After Pituitary Surgery)
Acronym: DHAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-05023
Record Dates: First submitted 2018-08-01; First posted 2018-08-17 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hyponatremia; Hyponatremic; Pituitary Tumor; Pituitary; Surgery
Keywords: hyponatremia; hyponatremic; pituitary tumor; transsphenoidal resection; pituitary surgery; pituitary
MeSH Terms: conditions — Hyponatremia; Pituitary Neoplasms; Pituitary Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Fluid restricted (Experimental): Fluids will be stopped at 8am on POD 1 and patients will be started on a moderate fluid restriction on POD #3 based on their weight (1000 cc/24 hours for patients who weigh <=100 kg and 1200 cc/24 hours for patients who weigh > 100kg)
  Interventions: Other: Fluid Restricted Group
- Non Fluid Restricted (No Intervention): No fluid restriction

INTERVENTIONS:
Other: Fluid Restricted Group — Patients will be started on a weight-based intravenous fluid replacement with D5 ½ NS on POD 0 (75 cc/hr for patients < 70kg, 100 cc/hr for patients 70-100kg, and 125 cc/hr for patients >100kg). Patients will be allowed to drink water freely after surgery on POD #0. Fluids will be stopped at 8am on POD 1 and patients will be started on a moderate fluid restriction on POD #3 based on their weight (1000 cc/24 hours for patients who weigh <=100 kg and 1200 cc/24 hours for patients who weigh > 100kg). Prior to initiation of a fluid restriction all of the following criteria have to be met:
  1. Serum Na level must be < 145 mEq/l
  2. Patient should be taking fluids by mouth
  3. Patient should not have evidence of DI (as determined by endocrine team following patient) If a patient in Fluid Restricted group develops DI, the fluid restriction will be stopped/not initiated.
  Arms: Fluid restricted

SUMMARY:
Hyponatremia is defined as sodium below the normal range of 135-145. Symptomatically, it can cause patients to experience a wide range of symptoms including lethargy, headache, nausea, vomiting and in severe cases coma and even death. The goal of this study is to prospectively compare two approaches to the postoperative fluid management of patients undergoing transsphenoidal resection of a pituitary tumor or cyst to decrease the occurrence of postoperative delayed hyponatremia. One group will be placed on moderate fluid restriction and the other group will be placed on ad lib fluid intake.

DETAILED DESCRIPTION:
Any adult patient with a pituitary adenoma (either non-functioning, prolactin-secreting, growth hormone secreting, gonadotropin secreting, or TSH (thyroid stimulating hormone) secreting) or cyst scheduled to undergo transsphenoidal resection will be included in the study. Patients with chronic hyponatremia will be excluded.

Patients will be randomly assigned to one of two groups:

Group 1: these patients will be treated with moderate fluid restriction (1000 ml/24 hours for patients <100kg and 1200 ml of fluid/24 hours for >100 kg starting on postoperative day 1. Fluid restriction will be aborted if diabetes insipidus occurs. Diabetes insipidus occurs if a patient does not produce enough ADH (anti-diuretic hormone) which is needed to concentrate the urine. Diabetes insipidus causes increased urination and increased thirst and can cause hypernatremia (an increased sodium level). A person will be diagnosed with diabetes insipidus if they meet all of the following criteria: serum sodium level > 146, dilute urine with a urine specific gravity < 1.003 and increased urine output defined by urine output > 300cc/hour for 2 consecutive hours( or > 6 liter/24 hours).

Group 2: these patients will not be placed on fluid restriction, they will be allowed to drink water freely after surgery.

All patients will be started on D5 ½ normal saline IV fluids (Weight based) and will be allowed to eat and drink starting on POD 1.

All the patients will receive a thirst questionnaire that will be completed daily starting on POD 1 until POD 13. The intensity of thirst will be assessed on a scale of 1--10, with 1 being no thirst, 5 being normal thirst and 10 being unbearable thirst.

Patients will have basic metabolic panels checked on post-surgical days 1, 3, 7, 10 and 13.

ELIGIBILITY:
Inclusion Criteria:

• Any adult patient with a pituitary adenoma or cyst (either non-functioning, prolactin-secreting, growth hormone secreting, ACTH (adrenocorticotropic hormone)-secreting, gonadotropin secreting, or TSH secreting) scheduled to undergo pituitary resection.

Exclusion Criteria:

* Patients with a history of chronic hyponatremia
* Patients with a history of SIADH (syndrome of inappropriate antidiuretic hormone) , except if secondary to hypothyroidism or adrenal insufficiency, or in association with prior TSS
* Patients with diabetes insipidus or patients receiving DDAVP
* Patients without an intact thirst mechanism
* Patients with CKD (chronic kidney disease) stage III, IV or V
* Patients with untreated adrenal insufficiency or hypothyroidism
* Patients with class III or IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Development of hyponatremia or low sodium | 3-14 days after surgery
  Sodium level <135 mEq/L

CONTACTS AND LOCATIONS:
Overall Officials: Julie Silverstein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Klaassen D, Mok S, Hwang JY, Blount SL, Williams KJ, Fong BM, Chicoine MR, Dacey RG, Farrell NF, Osbun JW, Rich KM, Roland LT, Schneider JS, Zipfel GJ, Luo C, Kim AH, Silverstein JM. Postoperative fluid restriction to prevent delayed hyponatremia after endoscopic transsphenoidal surgery. Neuro Oncol. 2025 Sep 8;27(7):1746-1757. doi: 10.1093/neuonc/noaf069. PMID 40084913